CLINICAL TRIAL: NCT06611423
Title: A Phase Ib, Double-blind, Placebo-controlled, Randomised Trial Investigating the Effect of AZD3427 on Renal Perfusion in HFrEF Patients With Renal Impairment Using Positron Emission Tomography (PET)
Brief Title: AZD3427 Effects on Renal Perfusion in Heart Failure Patients With Reduced Ejection Fraction and Renal Impairment
Acronym: Re-PERFUSE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor encountered difficulties in recruiting patients for clinical trial D8330C00004 and decided to end the study earlier for business reasons not affecting the benefit-risk balance.
Sponsor: AstraZeneca (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8330C00004
Record Dates: First submitted 2024-09-06; First posted 2024-09-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Renal Impairment
Keywords: Heart failure with reduced ejection fraction; HFrEF; Renal impairment; Reduced eGFR; AZD3427; PET
MeSH Terms: conditions — Renal Insufficiency | interventions — Dopamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IV Saline placebo followed by SC AZD3427 (Experimental): Participants will receive IV administration of saline only placebo prior to a PET examination. This is followed by a single SC dose of AZD3427 on Day 1 (V2).
  Interventions: Biological: AZD3427; Other: Radiolabelled ligand; Other: Saline
- IV Saline placebo followed by SC AZD3427 placebo (Placebo Comparator): Participants will receive IV administration of saline only placebo prior to a PET examination. This is followed by a single SC dose of AZD3427 Placebo on Day 1 (V2).
  Interventions: Other: AZD3427 Placebo; Other: Radiolabelled ligand; Other: Saline
- IV Dopamine diluted in saline followed by SC AZD3427 (Experimental): Participants will receive IV administration of dopamine diluted in saline prior to a PET examination. This is followed by a single SC dose of AZD3427 on Day 1 (V2)
  Interventions: Biological: AZD3427; Drug: Dopamine; Other: Radiolabelled ligand
- IV Dopamine diluted in saline followed by SC AZD3427 placebo (Placebo Comparator): Participants will receive IV administration of dopamine diluted in saline prior to a PET examination. This is followed by a single SC dose of AZD3427 Placebo on Day 1 (V2).
  Interventions: Other: AZD3427 Placebo; Drug: Dopamine; Other: Radiolabelled ligand

INTERVENTIONS:
Biological: AZD3427 — AZD3427 SC injection to be prepared using AZD3427 diluent
  Arms: IV Dopamine diluted in saline followed by SC AZD3427; IV Saline placebo followed by SC AZD3427
Other: AZD3427 Placebo — AZD3427 Placebo
  Arms: IV Dopamine diluted in saline followed by SC AZD3427 placebo; IV Saline placebo followed by SC AZD3427 placebo
Drug: Dopamine — Dopamine Hydrochloride 50mg/5mL
  Arms: IV Dopamine diluted in saline followed by SC AZD3427; IV Dopamine diluted in saline followed by SC AZD3427 placebo
Other: Radiolabelled ligand — Injection of radioligand for PET examinations
Other: Saline — Saline solution
  Arms: IV Saline placebo followed by SC AZD3427; IV Saline placebo followed by SC AZD3427 placebo

SUMMARY:
The present study is designed to test the effect of AZD3427 on renal perfusion in participants with heart failure and reduced eGFR (30 to 90 mL/min/1.73m2).

DETAILED DESCRIPTION:
This is a Phase Ib randomised, double-blind, placebo-controlled, single-dose, single-centre study to evaluate the renal haemodynamic effects of AZD3427 in participants with heart failure and reduced eGFR. This study will evaluate changes in the volumetric fraction of perfused renal cortex after a single dose of AZD3427 or AZD3427 placebo. These changes will be assessed using [15O]H2O PET imaging of the kidneys. Additional endpoints include changes in total renal perfusion, plasma/serum biomarkers of renal function, and safety and tolerability. Infusion with 2 to 4 µg/kg/min dopamine/saline placebo will be used as a positive control.

Study details include:

* The study duration will be up to 83 days.
* The treatment duration will be 1 day.
* The visit frequency will be on Day 1, Day 8 (± 3 days), and Day 56 (± 3 days).

ELIGIBILITY:
Inclusion Criteria

AGE:

- Participant must be > 20 years-old at the time of signing the informed consent.

DISEASE CHARACTERISTICS:

* Participant must have suitable veins for cannulation.
* Participants must have a known clinical diagnosis of HF NYHA I to III for at least 12 months.
* Participants must be on stable HF standard of care medication for at least 4 weeks prior to screening, with no significant dose change or new medications added during that period. If the participant is currently taking diuretics, then diuretics must also be stable for at least 4 weeks prior to screening. It is also expected that there will be no change in treatment between screening (Visit 1) and Visit 3 in terms of drugs known to affect renal haemodynamics, including but not limited to: ACE-Is, angiotensin II receptor blockers, angiotensin receptor-neprilysin inhibitors, mineralocorticoid receptor antagonists, cyclooxygenase inhibitors, endothelin receptors antagonists, phosphodiesterase inhibitors, SGLT2is, and diuretics.
* Participants must have a left ventricular ejection fraction of ≤ 40% based on echocardiography conducted within the last 6 months.
* Participants must have an eGFR of 30 to 90 mL/min/1.73 m2 (inclusive) assessed by the CKD-EPI, 2021 (creatinine only) equation without including race (Inker et al 2021) at screening.

BMI AND WEIGHT:

- Participants must have a minimum BMI of 18.0 kg/m2 and a minimum body weight of 50 kg at screening.

SEX AND CONTRACEPTIVE REQUIREMENTS:

* For female participants, the participant must not be pregnant or lactating and must be of non-childbearing potential, confirmed at screening by one of the following:

  1. Postmenopausal, defined as amenorrhoea for ≥ 12 months following cessation of all exogenous hormonal treatments, and with FSH levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not considered as irreversible surgical sterilisation.
* All male participants should refrain from fathering a child or donating sperm until 3 months after dosing. The female partner has to be either of non-childbearing potential or has to use a highly effective contraception form of birth control until 3 months after dosing. The female partner should be stable on their chosen method of birth control for at least 3 months prior to dosing.
* Male participants who have been sterilised are required to use one barrier method of contraception (condom) from the time of study intervention administration until 3 months after the dosing. The participant must have received medical assessment of the surgical success.

INFORMED CONSENT:

- Capable of and willing to give signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

MEDICAL CONDITIONS:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of screening or planned surgical or other procedure before study completion.
* Clinically significant, as judged by the investigator, ventricular arrhythmias requiring pharmacological treatment.
* Historical or current evidence of a clinically significant disease or disorder including, but not limited to:

  1. Myocardial infarction, stroke, transient ischaemic attack, coronary artery bypass grafting, percutaneous coronary intervention, implantable cardioverter defibrillator implantation, within 12 weeks prior to screening.
  2. Primary cardiomyopathy other than dilated, including but not limited to sarcoidosis, amyloidosis, restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy, complex congenital heart disease.
* Decompensated HF or hospitalisation due to any cause < 4 weeks prior to screening.
* Severe heart valve disease.
* Diagnosis of polycystic kidney disease or anatomical causes of chronic kidney disease.
* One kidney, renal artery stenosis, or glomerulonephritis.
* Anticipated dialysis or renal transplantation within 1 year.
* Condition where vasodilatory therapy maybe contraindicated for example but not limited to severe aortic stenosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy.
* History of active malignancy within 2 years, with the exception of fully excised or treated basal cell carcinoma or ≤ 2 squamous cell carcinomas of the skin.
* Participants who are under investigation for breast or cervical cancer, including participants with a pap smear of ≥ 3. All investigations must be resolved as negative for breast and cervical cancer at least 12 weeks before screening.
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator.
* Known or suspected history of drug abuse as judged by the Investigator.
* History of alcohol abuse or excessive intake of alcohol as judged by the Investigator, within the 6 months prior to screening.
* History of hypersensitivity to injection devices or to drugs with a similar chemical structure or class to AZD3427 or any component of the AZD3427 preparation, or to dopamine or any component of the dopamine preparation, or ongoing clinically important allergy/hypersensitivity.
* Participants who cannot communicate reliably with the Investigator.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Known history of ADAs to relaxin or relaxin analogues.
* Active infections that significantly affect the patient's health status or in the opinion of the Investigator, may put the participant at risk (eg, HIV, Hepatitis, tuberculosis, etc.).
* Plasma donation within 1 month prior to screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.

PRIOR/CONCOMITANT THERAPY:

- If on treatment with other drugs with potential to significantly influence on eGFR (eg, SGLT2i, ACE-I), the participant must have been on a stable dose for at least 4 weeks prior to screening.

PDE-5 inhibitors such as sildenafil (eg, taken for erectile dysfunction or other as-needed reasons) and NSAIDs such as diclofenac and ibuprofen should not be taken for 2 days before the PET Sessions 2 and 3 (Visit 2 and Visit 3); paracetamol is allowed.

PRIOR/CONCURRENT CLINICAL STUDY EXPERIENCE:

- Currently participating in or previous participation in another clinical study within 30 days prior to the Screening Visit or previous participation in another PET imaging trial within the last 12 months, or planned participation in such study prior to end of the Follow-up period.

Note: Participants consented and screened, but not entered in this study or a previous study, are not excluded.

DIAGNOSTIC ASSESSMENTS:

* Haemoglobin < 100 g/L at Screening.
* Abnormal vital signs defined as any of the following at screening:

  1. Sitting SBP > 160 mmHg or sitting DBP > 110 mmHg after a period of at least 5 minutes of rest;
  2. Sitting SBP < 100 mmHg or sitting DBP < 50 mmHg;
  3. Resting pulse rate of < 50 bpm or > 115 bpm.

OTHER EXCLUSIONS:

* Involvement of any AstraZeneca, CRO, or study centre employee or their close relatives, including any involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgement by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Previous enrolment or randomisation in the present study.
* For females only: currently pregnant (confirmed with positive pregnancy test) or breast-feeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
The volumetric fraction (%) of the renal cortex with increased perfusion from baseline to Day 8, compared to placebo. | Baseline to Day 8
  A PET image analysis of renal cortex measures the perfusion in approximately 8000 voxels. The volumetric fraction (%) is the fraction of voxels (%) with a positive change, i.e. increased perfusion.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Baseline to Day 56
  Number of participants with adverse events with onset after dose.
Number of participants with abnormal vital signs | Baseline to Day 56
  Predefined criteria for treatment-emergent changes in vital sign parameters will be used.
Number of participants with abnormal laboratory tests results | Baseline to Day 56
  Predefined criteria for treatment-emergent changes in laboratory parameters will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Azizi, MD, Principal Investigator — Clinical Trial Consultants
Locations (1):
- Research Site, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: ICF
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home